CLINICAL TRIAL: NCT05183256
Title: Development of the Cohort of the Patients With Inflammatory Bowel Disease in Yeouido St. Mary's Hospital
Brief Title: Cohort of Inflammatory Bowel Disease Patient in Yeouido St. Mary's Hospital
Status: Completed | Type: Observational
Sponsor: Yeouido St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Ilsoo Kim, MD, Principal Investigator, Yeouido St. Mary's Hospital
Other Study IDs: SC20TISI0103
Record Dates: First submitted 2021-12-01; First posted 2022-01-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples are collected to assess the severity of IBD. Tissue samples through colonoscopy biopsy and stool samples are collected to find out gut flora through DNA analysis. No human DNA analysis is targeted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pathologically Inflammatory bowel disease (IBD) is in chronic complex inflammatory gut pathological condition. Although the etiology of IBD is unknown, gut microbiota alteration (dysbiosis) is considered a novel factor involved in the pathogenesis of IBD. The aim of this study is to analyze gut microbiota in IBD patients.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) (Crohn's disease (CD) and ulcerative colitis (UC)) occurs worldwide with differences in epidemiology, etiology, and phenotype between regions. Pathologically Inflammatory bowel disease (IBD) is in chronic complex inflammatory gut pathological condition. Although the etiology of IBD is unknown, gut microbiota alteration (dysbiosis) is considered a novel factor involved in the pathogenesis of IBD. The DNA of microbiota will be investigated with samples of stool, colon tissue. The aim is to establish a cohort group for IBD (1), to make a database on cohort group characteristics such as endoscopic findings, disease severity, epidemiology, and prognosis (2), to analyze gut flora in IBD patients (3).

ELIGIBILITY:
Inclusion Criteria:

* The below 3 conditions must be met simultaneously.

  1. Patient who can voluntarily consent to this study.
  2. Patient who has inflammatory bowel disease.
  3. Patient who is aged less than 75 years.

Exclusion Criteria:

* a patient meets any of the below conditions.

  1. If a patient has an IBD other than UC and CD.
  2. If a patient is vulnerable due to his/her position as an employee of Yeouido St.Mary's hospital or a medical student of the Catholic University of Korea.
  3. If a patient is pregnant.
  4. Foreign personal who cannot speak Korean.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients with IBD, presented to division of gastroenterology, Yeouido St.Mary's hospital, will be asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with the remission of disease activity. | through study completion, an average of 2 year
  Disease activity is assessed in a clinical, endoscopic, and biochemical way. Each activity is determined by the Mayo score (in UC), Crohn's Disease Activity Index (in CD), Ulcerative Colitis Endoscopic Index of Severity (in UC), Simple Endoscopic Score for Crohn Disease (in CD), and biochemical findings (e.g. fecal calprotectin).

CONTACTS AND LOCATIONS:
Overall Officials: Ilsoo Kim, MD, Principal Investigator — Yeouido St. Mary's Hospital
Locations (1):
- Yeouido St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park SH, Kim YJ, Rhee KH, Kim YH, Hong SN, Kim KH, Seo SI, Cha JM, Park SY, Jeong SK, Lee JH, Park H, Kim JS, Im JP, Yoon H, Kim SH, Jang J, Kim JH, Suh SO, Kim YK, Ye BD, Yang SK; Songpa-Kangdong Inflammatory Bowel Disease [SK-IBD] Study Group. A 30-year Trend Analysis in the Epidemiology of Inflammatory Bowel Disease in the Songpa-Kangdong District of Seoul, Korea in 1986-2015. J Crohns Colitis. 2019 Oct 28;13(11):1410-1417. doi: 10.1093/ecco-jcc/jjz081. PMID 30989166
- [Result] Dalal SR, Chang EB. The microbial basis of inflammatory bowel diseases. J Clin Invest. 2014 Oct;124(10):4190-6. doi: 10.1172/JCI72330. Epub 2014 Aug 1. PMID 25083986